CLINICAL TRIAL: NCT03987412
Title: Diabetes Mellitus, Impaired Glucose Tolerance and Gestational Diabetes Mellitus Intervention Action-Leading Trial- Gestational Diabetes Mellitus Study
Brief Title: A Behavioral Intervention to Prevent Gestational Diabetes Mellitus
Acronym: DIGITAL-G
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DIGITAL-G-2019
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-04

CONDITIONS: Diabetes, Gestational
Keywords: Behavioral intervention; First trimester; Gestational diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral intervention (Experimental): Pregnant women randomized to the behavioral intervention group will recieve a face-to-face education about the risks of GDM at their local rearch centers. Then they will be provided with a mobile APP incorporating nutrition, exercise and phycological support. They will also have regular prenatal care in their local hospitals.
  Interventions: Behavioral: Lifestyle intervention with APP
- Control group (No Intervention): Pregnant women randomized to the control group only have regular prenatal care in their local hospitals.

INTERVENTIONS:
Behavioral: Lifestyle intervention with APP — The face to face education class will be conducted by an obstetrician, an endocrinologist and a nutritionist together. Then the lifestyle intervention will be launched by an APP that installed in participants' private mobile phones, including nutrition, exercise and phycological support. Nutrition guidance is conducted according to the Chinese Dietary Guide, Chinese and international guidelines of gestation diabetes management. Exercise support is given based on the Guidelines for National Fitness of China, Chinese and international guidelines of gestation diabetes. Phycological support is given by sending education articles on mental health. Participants are encouraged to update data about their diet, exercise and body weight through the APP, and based on the data investigators will individualize the suggestions.
  Arms: Behavioral intervention

SUMMARY:
Gestational diabetes mellitus (GDM) increases the risk of adverse pregnancy outcome and developing type 2 diabetes after delivery. It is well recognized that behavioral intervention is effective in preventing type 2 diabetes in high risk population. Recently, some studies showed that exercise, dietary and weight control reduced the risk of developing GDM in obese/over weight women or in women with GDM history. With the increasing use of smartphones, mobile applications (APPs) can be applied in the education and management of chronic diseases, including diabetes. Therefore, the investigators will conduct a multi-centered, two-armed, open-labeled, randomized controlled trial to evaluate whether early lifestyle intervention with a mobile APP can prevent the occurrence of GDM in pregnant women who are at high risk of this disease.

The investigators hypothesis that behavioral intervention from the first trimester of pregnancy with mobile APP that incorporates nutrition, exercise and phycological support will:

1. Reduce the risk of developing GDM in pregnant women with risks of GDM.
2. Improve the pregnant women's adherence of behavioral intervention and their satisfaction of prenatal medical care.

DETAILED DESCRIPTION:
Participates will be recruited from five research centers in the mainland of China. Pregnant women will be screened for risks of GDM at their first visit for prenatal care during their first trimester (less than 12 gestational weeks). Obstetricians will introduce the study to women who have one or more risk factors.

Women who meet the eligibility criteria and who are willing to provide informed consent will be enrolled and randomized to behavioral intervention group and control group. Women in the behavioral intervention group will be educated about the risks of GDM, and then applied with a mobile APP that provides nutrition, exercise and phycological support starting from their first trimester. This behavioral support will be modified individually and continuously according to the pregnant women's feedback of their daily performance through the APP. Both groups will have regular prenatal care.

During 24-28 gestational weeks, GDM will be diagnosed by a 75g oral glucose tolerance test (OGTT) according to the new World Health Organization criteria as fasting glucose level in fasting whole blood ≥5.1mmol/L, or 1-hour value ≥10.0mmol/l, or 2-hour value ≥8.5mmol/L. Investigators will compare the GDM risk in the two groups to evaluate whether behavioral intervention with mobile APP can reduce the risk of GDM in Chinese pregnant women who are at high risk of GDM. Participants' adherence with the behavioral intervention will be evaluated by analyzing the data collected by the APP, and participants' satisfaction of the prenatal care will be evaluated with questionnaires during 24-28 gestational weeks. Intervention with the APP will be stopped in the third trimester. All the participates will receive standard medical management until they give birth.

ELIGIBILITY:
Inclusion Criteria:

* Chinese pregnant women aged between 30 and 45 years who have one or more risk factors when they are on their first prenatal care visit. The risk factors are listed as following:

  1. Fasting plasma glucose level ≥ 4.4 mmol/l.
  2. Body mass index ≥ 24 kg/m^2
  3. Systolic blood pressure ≥ 130 mmHg, or diastolic blood pressure ≥ 80 mmHg.
  4. First-degree family history of diabetes
  5. History of GDM
  6. History of polycystic ovary syndrome.
* Willing to keep reading the education articles and supporting materials that delivered by the mobile APP.
* Willing to provide informed consent.

Exclusion Criteria:

* First prenatal care visit later than 12 gestational weeks
* Fasting plasma glucose level value ≥5.6 mmol/l, or glycated hemoglobin value ≥ 5.6%.
* Continuous use of antidiabetic medicine for 7 days or more within the current 3 months
* Spontaneous abortion twice or more
* Body weight loss for 10% or more within the current 3 months
* History of other diseases including but not limited to:

  1. Arteriosclerotic cardiovascular disease, heart failure or stroke
  2. Systolic blood pressure ≥160 mmHg, or diastolic blood pressure ≥90 mmHg.
  3. Hematological system diseases. For anemia patients, hemoglobin ≥90g/l is acceptable.
  4. Renal dysfunction or liver dysfunction
  5. Rheumatic diseases, currently receiving glucocorticoids or other immunosuppressors
  6. Serious diseases of respiratory system with current use of glucocorticoids.
  7. Diseases of endocrine system. But it is acceptable that the hypothyroidism has been controlled with levothyroxine.
* Other conditions that investigators consider inappropriate for this study.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The risk of gestational diabetes mellitus (GDM) | 24-28 gestational weeks
  GDM will be diagnosed by a 75g OGTT according to the World Health Organization criteria as fasting plasma glucose level ≥5.1 mmol/L, or 1-hour value ≥10.0mmol/l, or 2-hour value ≥8.5mmol/L. Investigators will calculate the occurrence rate of GDM to represent the risk of GDM.

SECONDARY OUTCOMES:
Adherence of behavioral intervention during pregnancy | up to 28 gestational weeks
  Participants will be encouraged to update their data about their diet, exercise and body weight. The frequency of their update and feedback data will be used to evaluate the adherence of behavioral intervention.
Satisfaction of prenatal medical care; questionnaires | up to 24-28 gestational weeks
  Participants' satisfaction of prenatal medical care will be evaluated with questionnaires. The questionnaire was designed by the investigators according to references (Stoyanov SR. JMIR Mhealth Uhealth, 2015, 1(3): e27. et al) named the " Satisfaction Questionnaire of Behavioral Intervention to Prevent GDM". It includes 7 subscales. The final form of each subscale is a five-point scale (5 Strongly agree / 4 agree / 3 don't know / 2 disagree / 1 strongly disagree, modified from Likert Scale) which is used to allow the participants to express how much they agree or disagree with the satisfaction statement.
  1. Convenience and feasibility of behavioral intervention
  2. Effects of behavioral intervention
  3. Behavioral intervention do not have adverse reactions
  4. Ease use of APP
  5. Good engagement of APP
  6. High information quality of APP
  7. The investigators serve well
  Summarize each scale to compute a total score. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Tianpei, MD,PhD, Principal Investigator — Department of Endocrinology and Metabolism, Peking University Third Hospital
Locations (1):
- Haidian Maternal&Child Health Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No